CLINICAL TRIAL: NCT04213209
Title: Special Drug Use Surveillance for Adcetris Intravenous Infusion 50 Milligrams "Relapsed or Refractory CD30-positive Peripheral T Cell Lymphoma or Hodgkin Lymphoma (Only Pediatric Patients)"
Brief Title: Special Drug Use Surveillance for Brentuximab Vedotin Intravenous Infusion "Relapsed or Refractory CD30-positive Peripheral T Cell Lymphoma or Pediatric Hodgkin Lymphoma"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C25021; jRCT1080224999 (Registry Identifier: jRCT)
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-06

CONDITIONS: Peripheral T Cell Lymphoma; Pediatric Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Brentuximab Vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brentuximab Vedotin 1.8 mg/kg (body weight): The usual dosage for intravenous administration is 1.8 milligrams per kilograms (mg/kg) (body weight) as Brentuximab Vedotin (genetic recombination) once every three weeks (up to 12 months). The dose may be reduced appropriately according to the participant's condition. Participants receive interventions as part of routine medical care.
  Interventions: Drug: Brentuximab Vedotin (Genetical Recombination)

INTERVENTIONS:
Drug: Brentuximab Vedotin (Genetical Recombination) — Brentuximab Vedotin Intravenous Infusion
  Other Names: ADCETRIS Intravenous Infusion 50 mg

SUMMARY:
The purpose of this survey is to examine the safety of adult patients with relapsed or refractory CD30-positive peripheral T-cell lymphoma (PTCL) (excluding anaplastic large cell lymphoma (ALCL)) and pediatric patients with relapsed or refractory CD30-positive PTCL or Hodgkin lymphoma (HL) in the actual use of on concomitant Brentuximab Vedotin in routine clinical practice.

DETAILED DESCRIPTION:
The drug being tested in this survey is called Brentuximab Vedotin intravenous infusion 50 mg. This intravenous infusion is being tested to treat adult patients with relapsed or refractory CD30-positive peripheral T-cell lymphoma (PTCL) (excluding anaplastic large cell lymphoma (ALCL)) and pediatric patients with relapsed or refractory CD30-positive PTCL or Hodgkin lymphoma (HL).

This survey is an observational (non-interventional) study and will look at the safety of adult patients with relapsed or refractory CD30-positive PTCL (excluding ALCL) and pediatric patients with relapsed or refractory CD30-positive PTCL or HL in the routine clinical setting. The number of observed patients will be approximately 86 as total (80; Adult participants and 6; Pediatric participants).

This multi-center observational survey will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with relapsed or refractory lymphoma.
2. CD30-positive participants.
3. Participants who receive study drug after obtaining approval of CD30-positive PTCL indication of study drug.

Exclusion Criteria:

1. Participants with a history of severe hypersensitivity to Brentuximab Vedotin.
2. Participants taking bleomycin hydrochloride treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with relapsed or refractory CD30-positive PTCL (excluding ALCL) and pediatric patients with relapsed or refractory CD30-positive PTCL or HL as part of routine medical care.
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a36e

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 50 investigative sites in Japan, from 14 February 2020 to 13 December 2023.
Pre-assignment Details: Adult participants with a historical diagnosis of relapsed or refractory CD30-positive peripheral T-cell lymphoma (PTCL) (excluding anaplastic large cell lymphoma (ALCL)) and pediatric participants with a historical diagnosis of relapsed or refractory CD30-positive PTCL or Hodgkin lymphoma (HL) were enrolled. Participants received Brentuximab Vedotin Intravenous Infusion as part of a routine medical care.
Groups:
- Adult Participants With PTCL-NOS: Adult participants with peripheral T-cell lymphoma not otherwise specified (PTCL-NOS) were received brentuximab vedotin (genetic recombination) 1.8 milligrams per kilograms (mg/kg) (body weight), intravenous infusion, once every three weeks (up to 12 months). The dose should be reduced appropriately depend on the participant's condition. Participants received interventions as part of routine medical care.
- Adult Participants With AITL: Adult participants with angioimmunoblastic T-cell lymphoma (AITL) were received brentuximab vedotin (genetic recombination) 1.8 milligrams per kilograms (mg/kg) (body weight), intravenous infusion, once every three weeks (up to 12 months). The dose should be reduced appropriately depend on the participant's condition. Participants received interventions as part of routine medical care.
- Adult Participants With ATLL: Adult participants with adult T-cell leukemia/lymphoma (ATLL) were received brentuximab vedotin (genetic recombination) 1.8 milligrams per kilograms (mg/kg) (body weight), intravenous infusion, once every three weeks (up to 12 months). The dose should be reduced appropriately depend on the participant's condition. Participants received interventions as part of routine medical care.
- Adult Participants With Other PTCL: Adult participants with the other PTCL (peripheral T-cell lymphoma [PTCL] subtypes other than anaplastic large-cell lymphoma [ALCL] [not surveyed], PTCL-NOS, AITL, and ATLL) were received brentuximab vedotin (genetic recombination) 1.8 milligrams per kilograms (mg/kg) (body weight), intravenous infusion, once every three weeks (up to 12 months). The dose should be reduced appropriately depend on the participant's condition. Participants received interventions as part of routine medical care.
- Pediatric Participants With PTCL: Pediatric participants with peripheral T-cell lymphoma (PTCL) were received brentuximab vedotin (genetic recombination) 1.8 milligrams per kilograms (mg/kg) (body weight), intravenous infusion, once every three weeks (up to 12 months). The dose should be reduced appropriately depend on the participant's condition. Participants received interventions as part of routine medical care.
- Pediatric Participants With HL: Pediatric participants with Hodgkin lymphoma (HL) were received brentuximab vedotin (genetic recombination) 1.8 milligrams per kilograms (mg/kg) (body weight), intravenous infusion, once every three weeks (up to 12 months). The dose should be reduced appropriately depend on the participant's condition. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
Started | 32 | 35 | 14 | 6 | 4 | 4
Completed | 31 | 35 | 14 | 6 | 4 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL | Total
Number analyzed (Participants) | 31 | 35 | 14 | 6 | 4 | 4 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.9 (12.01) | 72.6 (9.23) | 68.0 (12.82) | 49.2 (23.52) | 12.3 (3.69) | 12.0 (4.24) | 64.4 (20.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 9 | 4 | 1 | 2 | 48
  Male | 18 | 16 | 5 | 2 | 3 | 2 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 31 | 35 | 14 | 6 | 4 | 4 | 94
Duration of Diagnosis of PTCL or HL [Mean (Standard Deviation); unit: Months] — Mean duration between the first diagnosis of relapsed or refractory CD30 positive peripheral T-cell lymphoma (PTCL) or Hodgkin lymphoma (HL: pediatric participants only) and the first dose was reported.
  Months | 35.7 (42.96) | 31.0 (36.30) | 37.2 (64.90) | 5.7 (8.57) | 5.0 (2.94) | 18.3 (12.69) | 30.2 (42.01)
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance status assess participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than [>] 50 percent [%] of waking hours), capable of all self-care, unable to carry out any work activities; 3=capable of only limited selfcare, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5=dead.
  Participants
    Scale = 0 | 11 | 11 | 5 | 3 | 1 | 4 | 35
    Scale = 1 | 13 | 17 | 6 | 3 | 2 | 0 | 41
    Scale = 2 | 5 | 5 | 1 | 0 | 0 | 0 | 11
    Scale = 3 | 1 | 1 | 2 | 0 | 1 | 0 | 5
    Scale = 4 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Healthcare Category [Count of Participants; unit: Participants]
  Outpatient | 7 | 2 | 3 | 1 | 0 | 2 | 15
  Inpatient | 24 | 33 | 11 | 5 | 4 | 2 | 79
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 11 | 8 | 6 | 1 | 2 | 2 | 30
    Had Medical Complications | 20 | 27 | 8 | 5 | 2 | 2 | 64
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above. Unknown: Data could not be collected.
  Participants
    Had No Medical History | 18 | 21 | 11 | 4 | 4 | 3 | 61
    Had Medical History | 13 | 13 | 3 | 2 | 0 | 1 | 32
    Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 1
Smoking Classification [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Never Smoked | 12 | 14 | 6 | 4 | 4 | 4 | 44
    Current Smoker | 1 | 3 | 0 | 1 | 0 | 0 | 5
    Ex-Smoker | 12 | 9 | 7 | 1 | 0 | 0 | 29
    Unknown | 6 | 9 | 1 | 0 | 0 | 0 | 16
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 57.65 (11.031) | 54.01 (12.328) | 52.14 (10.082) | 56.77 (12.517) | 41.75 (7.677) | 47.00 (21.386) | 54.29 (12.167)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2]
  Kilogram (kg)/meter (m)^2 | 22.20 (3.536) | 21.85 (3.764) | 20.86 (4.059) | 22.43 (5.033) | 18.08 (2.981) | 20.73 (5.239) | 21.65 (3.858)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Serious or Non-serious Adverse Event Classified as Peripheral Neuropathy
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Percentage of participants who had one or more serious or non-serious adverse event of peripheral motor neuropathy or peripheral sensory neuropathy which were classified as peripheral neuropathy was reported.
Time Frame: Up to 12 Months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
Number analyzed (Participants) | 31 | 35 | 14 | 6 | 4 | 4
Participants
  Serious: Peripheral Motor Neuropathy | 0 | 0 | 0 | 0 | 0 | 0
  Non-Serious: Peripheral Motor Neuropathy | 1 | 0 | 0 | 1 | 0 | 0
  Serious: Peripheral Sensory Neuropathy | 0 | 1 | 0 | 0 | 0 | 0
  Non-Serious: Peripheral Sensory Neuropathy | 8 | 9 | 2 | 1 | 2 | 0

2. Primary Outcome: Percentage of Participants Who Had One or More Serious or Non-serious Adverse Drug Reaction Classified as Peripheral Neuropathy
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug. Percentage of participants who had one or more serious or non-serious adverse drug reaction of peripheral motor neuropathy or peripheral sensory neuropathy which were classified as peripheral neuropathy was reported.
Time Frame: Up to 12 Months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
Number analyzed (Participants) | 31 | 35 | 14 | 6 | 4 | 4
Participants
  Serious: Peripheral Motor Neuropathy | 0 | 0 | 0 | 0 | 0 | 0
  Non-Serious: Peripheral Motor Neuropathy | 1 | 0 | 0 | 1 | 0 | 0
  Serious: Peripheral Sensory Neuropathy | 0 | 1 | 0 | 0 | 0 | 0
  Non-Serious: Peripheral Sensory Neuropathy | 8 | 9 | 2 | 1 | 2 | 0

3. Primary Outcome: Percentage of Participants Who Had One or More Serious or Non-serious Adverse Event Classified as Myelosuppression
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Percentage of participants who had one or more serious or non-serious adverse event of febrile neutropenia, neutropenia, or neutrophil count decreased which were classified as myelosuppression was reported.
Time Frame: Up to 12 Months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
Number analyzed (Participants) | 31 | 35 | 14 | 6 | 4 | 4
Participants
  Serious: Febrile Neutropenia | 1 | 1 | 0 | 0 | 1 | 0
  Non-Serious: Febrile Neutropenia | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Neutropenia | 1 | 0 | 0 | 0 | 1 | 0
  Non-Serious: Neutropenia | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Neutrophil Count Decreased | 3 | 0 | 0 | 0 | 0 | 0
  Non-Serious: Neutrophil Count Decreased | 9 | 3 | 2 | 0 | 0 | 1

4. Primary Outcome: Percentage of Participants Who Had One or More Serious or Non-serious Adverse Drug Reaction Classified as Myelosuppression
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug. Percentage of participants who had one or more serious or non-serious adverse drug reaction of febrile neutropenia, neutropenia, or neutrophil count decreased which were classified as myelosuppression was reported.
Time Frame: Up to 12 Months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
Number analyzed (Participants) | 31 | 35 | 14 | 6 | 4 | 4
Participants
  Serious: Febrile Neutropenia | 1 | 0 | 0 | 0 | 0 | 0
  Non-Serious: Febrile Neutropenia | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Neutropenia | 1 | 0 | 0 | 0 | 0 | 0
  Non-Serious: Neutropenia | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Neutrophil Count Decreased | 3 | 0 | 0 | 0 | 0 | 0
  Non-Serious: Neutrophil Count Decreased | 9 | 3 | 2 | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants Who Had One or More Serious or Non-serious Adverse Event Classified as Lung Disorder
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Percentage of participants who had one or more serious or non-serious adverse event of only interstitial lung disease which were classified as lung disorder was reported.
Time Frame: Up to 12 Months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
Number analyzed (Participants) | 31 | 35 | 14 | 6 | 4 | 4
Participants
  Serious: Interstitial Lung Disease | 1 | 1 | 0 | 0 | 0 | 0
  Non-Serious: Interstitial Lung Disease | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Percentage of Participants Who Had One or More Serious or Non-serious Adverse Drug Reaction Classified as Lung Disorder
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug. Percentage of participants who had one or more serious or non-serious adverse drug reaction of only interstitial lung disease which were classified as lung disorder was reported.
Time Frame: Up to 12 Months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
Number analyzed (Participants) | 31 | 35 | 14 | 6 | 4 | 4
Participants
  Serious: Interstitial Lung Disease | 1 | 1 | 0 | 0 | 0 | 0
  Non-Serious: Interstitial Lung Disease | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Who Achieve or Maintain Any Best Response for Adult Participants With PTCL-NOS, AITL, the Other PTCL, and Pediatric Participants With PTCL
Description: Best response is defined as the cumulative numbers of participants who achieve each level of best response including complete response (CR), complete response uncertain (CRu) (when no positron emission tomography [PET] data are available), partial response (PR), Stable Disease (SD), and Progressive Disease (PD) after treatment. Best response was assessed by the antitumor response criteria for adult PTCL. Reported data are divided into 2 populations; with or without PET data for each group. PET was used in cancer diagnosis and treatment.
Time Frame: Up to 12 Months
Population: Efficacy analysis set: all participants who received at least one dose of protocol treatment without major protocol deviation. The number analyzed was the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With Other PTCL | Pediatric Participants With PTCL
Number analyzed (Participants) | 24 | 27 | 3 | 1
Participants
  With PET Assessment: number analyzed (Participants) | 9 | 14 | 1 | 1
  With PET Assessment | 7 | 12 | 0 | 1
  Without PET Assessment: number analyzed (Participants) | 15 | 13 | 2 | 0
  Without PET Assessment | 4 | 5 | 0 | 0

8. Secondary Outcome: Percentage of Participants Who Achieve or Maintain Any Best Response for Adult Participants With ATLL
Description: Best response is defined as the cumulative numbers of participants who achieve each level of best response including complete response (CR), partial response (PR), Stable Disease (SD), and Progressive Disease (PD) after treatment. Best response was assessed by the antitumor response criteria.
Time Frame: Up to 12 Months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With ATLL
Number analyzed (Participants) | 11
Participants | 3

9. Secondary Outcome: Percentage of Participants Who Achieve or Maintain Any Best Response for Pediatric Participants With PTCL and HL
Description: Best response is defined as the cumulative numbers of participants who achieve each level of best response including complete response (CR), complete response uncertain (CRu) (for PTCL), partial response (PR), Stable Disease (SD), and Progressive Disease (PD) after treatment. Best response was assessed by the Japanese Pediatric Leukemia/Lymphoma Study Group (JPLSG) version of antitumor response criteria.
Time Frame: Up to 12 Months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Participants With PTCL | Pediatric Participants With HL
Number analyzed (Participants) | 3 | 3
Participants | 3 | 2

10. Secondary Outcome: Percentage of Participants Who Had One or More Adverse Event
Description: AE is defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Up to 12 Months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
Number analyzed (Participants) | 31 | 35 | 14 | 6 | 4 | 4
Participants | 21 | 22 | 8 | 5 | 3 | 3

11. Secondary Outcome: Percentage of Participants Who Had One or More Adverse Drug Reaction
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Up to 12 Months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
Number analyzed (Participants) | 31 | 35 | 14 | 6 | 4 | 4
Participants | 20 | 18 | 6 | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 12 Months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Adult Participants With PTCL-NOS | Adult Participants With AITL | Adult Participants With ATLL | Adult Participants With Other PTCL | Pediatric Participants With PTCL | Pediatric Participants With HL
All-Cause Mortality (participants affected / at risk) | 1/31 | 5/35 | 2/14 | 0/6 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 8/31 | 12/35 | 2/14 | 1/6 | 3/4 | 2/4
Other Adverse Events (participants affected / at risk) | 18/31 | 14/35 | 6/14 | 4/6 | 2/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Participants With PTCL-NOS (N=31) | Adult Participants With AITL (N=35) | Adult Participants With ATLL (N=14) | Adult Participants With Other PTCL (N=6) | Pediatric Participants With PTCL (N=4) | Pediatric Participants With HL (N=4)
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Angioimmunoblastic T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 0 | 0 | 0
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 4 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Participants With PTCL-NOS (N=31) | Adult Participants With AITL (N=35) | Adult Participants With ATLL (N=14) | Adult Participants With Other PTCL (N=6) | Pediatric Participants With PTCL (N=4) | Pediatric Participants With HL (N=4)
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 9 | 2 | 1 | 2 | 0
VIth nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 9 | 3 | 2 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT04213209/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT04213209/SAP_001.pdf